CLINICAL TRIAL: NCT06404697
Title: Evaluating the Efficacy and Safety of Boost Irradiation to the Supraclavicular Area Among High Risk cN3c Breast Cancer Patients According to Nodal Response: a Single-arm, Prospective Clinical Study
Brief Title: Boost Irradiation to the Supraclavicular Area Among High Risk cN3c Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuijinH 2024(026)
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: cN3c; Boost irradiation; breast cancer; high risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk (Experimental): High-risk patients will undergo boost irradiation to the SCV with a cumulative dose of ≥60 Gy.
  Interventions: Radiation: Boost irradiation

INTERVENTIONS:
Radiation: Boost irradiation — High-risk patients will undergo boost irradiation to the SCV with a cumulative dose of ≥60 Gy.

SUMMARY:
cN3c breast cancer with ipsilateral supraclavicular (SCV) lymph nodal (SCLN) metastasis is known to have a dismal prognosis. Currently, the combined-modality therapy consisting of primary systemic therapy (PST), subsequent local and/or systemic therapy based on response is the standard of care. However, the value of giving radiotherapy (RT) boost to SCV region remains uncertain in cN3c patients. This study aimed to assess the efficacy and safety of RT boost to the SCV area in high-risk cN3c breast cancer patients based on nodal response following PST.

DETAILED DESCRIPTION:
This study is a phase II single-arm, prospective clinical trial aimed at assessing the efficacy and safety of RT boost to the SCV area among high-risk cN3c breast cancer patients contingent upon the nodal response after PST.

Our previous retrospective study revealed that nodal response to PST serves as an independent prognostic factor for survival and pattern of failure. A cumulative SCV dose of ≥60 Gy has been associated with improved overall survival (OS) in subgroup of patients who did not achieve SCLN cCR.

Based on nodal response to PST, patients will be categorized into three groups: those who did not achieve cCR in SCLN (considered high risk), those who achieved SCLN cCR but did not attain pCR in ALN (considered intermediate risk), and those who achieved cCR in SCLN and pCR in ALN (considered low risk). High-risk patients will undergo boost irradiation to the SCV with a cumulative dose of ≥60 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation with documented informed consent.
* Females aged ≥18 years.
* Histological or cytological confirmed primary breast carcinoma.
* Clinical diagnosis of cN3c.
* Receipt of neoadjuvant therapy, guided by the attending physician and current treatment guidelines.
* Did not achieve cCR in SCLN following neoadjuvant therapy.
* Undergoing curative-intent breast cancer surgery post-neoadjuvant therapy.
* Pathological evaluation of axillary lymph nodes post-surgery.
* KPS score ≥80, with expected survival exceeding 2 years.
* Complete healing of surgical incision without complications.
* Negative pathological surgical margins.
* Availability of hormonal receptor (ER/PR), HER2, and Ki-67 status for the primary breast lesion.
* Pre-menopausal females required to practice contraception for at least one month prior to screening, maintaining contraception throughout the study and for a specified period post-study cessation.

Exclusion Criteria:

* Patients with confirmed distant metastases by pathology or imaging.
* Those who have not received neoadjuvant systemic therapy.
* Patients who have not undergone curative-intent surgery.
* Pregnant or lactating women.
* Individuals with severe non-neoplastic comorbidities affecting radiotherapy implementation.
* History of malignancy within the past 5 years (excluding ductal carcinoma in situ, basal cell carcinoma, squamous cell carcinoma in situ, cervical carcinoma in situ, and in situ adenocarcinoma of the lung).
* Simultaneous contralateral breast cancer.
* History of prior radiation therapy to the neck, chest, or ipsilateral axilla.
* Active collagen vascular disease.
* Patients with T4 staging of the primary tumor.
* Inability to initiate radiotherapy within 12 weeks post breast cancer curative surgery (breast-conserving surgery or mastectomy), or within 8 weeks post completion of adjuvant chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival | 2 years
  RFS were calculated from the date of surgery to the date of first documented recurrence (including regional, local and distant) or mortality, whichever happens first. In the case of patients who had not encountered recurrence or death, specifically in terms of recurrence-free survival, the time of the last tumor assessment was considered as the endpoint. Tumor response was evaluated by investigators following RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival | 2 years
  defined as the period from the initial drug administration to the subject's demise from various causes. In cases where patients were lost to follow-up prior to their passing, the date of their last documented contact was documented. For patients still alive at the last analyzed time point, the time of their last contact was considered as their survival duration. In the analysis of survival and subsequent treatment, all patients were monitored until their death, loss to follow-up, or the conclusion of the study.
Late toxicity | 2 years
  Monitor the occurrence of late toxic reactions (based on CTCAE 5.0) after 6 months after the completion of radiotherapy
Acute toxicity | 6 months
  Monitor the occurrence of acute toxic reactions (based on CTCAE 5.0) and subacute toxic reactions (RTOG) in the treatment of cN3c radiotherapy, both during the treatment course and within three months after its completion.
Quality of Life (QoL) | 2 years
  Collect QoL data on cN3c breast cancer patients. The data is measured by EORTC QLQ-C30 (Version 3.0) according to investigator collection at the starting and ending time of the treatment. EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The core and disease-specific for ESCC modules are selected to estimate treatment related influence on patients' life. The final score of the questionnaire is collected and analyzed according to detailed scoring procedures from manuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This is our retrospective study relevant to this trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10344941/